CLINICAL TRIAL: NCT00180843
Title: Assessment of Ventilation-perfusion Abnormalities in Patients With Smoking-related Airways Disease in Stable Condition and the Effect of Bronchodilator Therapy
Brief Title: Assessment of Ventilation-perfusion Abnormalities in Patients With Stable Smoking-related Airways Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of resources research fellow left
Sponsor: Imperial College London (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Philip Ind, Consultant Physician, Imperial College London
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 04/6741
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Ipratropium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- saline control (Placebo Comparator): nebulized saline
  Interventions: Drug: nebulized saline
- salbutamol and ipratropium bromide nebules (Active Comparator): salbutamol 2.5 mg and ipratropium bromide 0.5 mg
  Interventions: Drug: salbutamol + ipratropium bromide nebules

INTERVENTIONS:
Drug: salbutamol + ipratropium bromide nebules
  Other Names: albuterol; Ventolin; Atrovent
  Arms: salbutamol and ipratropium bromide nebules
Drug: nebulized saline
  Arms: saline control

SUMMARY:
Subjects undergo history, examination, lung function assessment after informed consent has been obtained. All subjects will undergo ventilation-perfusion scans. If there first scan is normal they will undergo a second and final scan four weeks later. If abnormal they will undergo two further scans with either nebulized bronchodilator or nebulized saline prior to their second and third scans. Each time they will have repeat lung function tests prior to scanning. We will examine the regional changes in ventilation and perfusion and there relationship to lung function.

DETAILED DESCRIPTION:
As in Brief description

ELIGIBILITY:
Inclusion Criteria:

* FEV1 < 70% predicted at baseline on spirometry
* significant smoking history or alpha 1 antitrypsin deficiency
* no evidence of current infection or restrictive lung disease

Exclusion Criteria:

* history of other significant respiratory disease
* significant respiratory infection within 6 weeks
* history of significant physical or mental illness rendering them unfit for the study in the opinion of the investigator
* taken part in any other research within the past 12 months, or received exposure to ionizing radiation

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
scan grade | post scan
  previously validated grading score

SECONDARY OUTCOMES:
lung function | pre scan

CONTACTS AND LOCATIONS:
Overall Officials: Philip W Ind, MB BChir MRCP, Principal Investigator — Imperial College Hammersmith
Locations (1):
- Imperial College Hammersmith Campus, London, London, United Kingdom